Dual-plane Ultrasound Imaging During Vascular Access Procedures

NCT05093699

September 1, 2023

## Statistical Analysis Plan

Quantitative, patient-outcomes:

Continuous outcome summarized using mean and category outcome summarized via frequency. Log transformation analysis used to satisfied distribution all assumptions. Assessed via on adjusted linear regression. Exploratory analysis. Statistical significance determined by two-tailed p-values of 0.05 or less. Data management and statistical analyses were performed in SAS 9.4

Qualitative, provider-response questions:

Theme based analysis utilizing verbatim responses. Assignment of code numbers to the themes and application two individual responses. Frequency of theme in total and subgroup analysis to be reported.